CLINICAL TRIAL: NCT06280404
Title: Body First Approach in Laparoscopic Cholecystectomy in Cases With Obscure Calot's Triangle
Brief Title: Body First Approach in Lap Cholecystectomy in Cases With Obscure Calot's Triangle
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Abdullah Badawy, Doctor, Assiut University
Other Study IDs: Body first in lap chole
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lap cholecystectomy — Body first approach in laparoscopic cholecystectomy in cases with obscure Calot's triangle

SUMMARY:
The aim of this study is to evaluate the body first approach on the rate of conversion to open technique & VBI in patients with obscure calot's triangle.

DETAILED DESCRIPTION:
Gallbladder disease is one of the most common reasons patients are referred to a general surgeon. Laparoscopic cholecystectomy (LC) is the current standard of care for symptomatic cholelithiasis. Despite being considered a low-risk surgery, bile duct injuries (BDIs) have occurred at a constant rate in the last 30 years, leaving devastating consequences on the affected patients. However vasculobiliary injury (VBI) is a rare but critical complication of (LC). So we need to follow critical view of safety. The critical view of safety (CVS) described by Strasberg is considered as the one of the most important critical factors for overall safety during LC. The CVS consists of three essential component or steps: 1) dissection of the hepatocystic triangle (HCT); 2) exposure of at least lower one third of the cystic plate (CP); and 3) demonstration of only two tubular structures (cystic duct and cystic artery) that remain attached to the gallbladder (after components 1 and 2 are achieved). All these three steps must be completed before considering that CVS has been achieved. However in some cases Calot's triangle can't be demonstrated due to dense adhesions. Conversion with retrograde approach (fundus first) was an option for these cases. However a retrograde approach can be achieved laparoscopically by starting dissection by body to use the fundus attachment for retraction which is called (the "body-first approach") that may decrease the possibility of VBI. Recent studies deficient in evaluation of outcome of (body first approach). So the interest of our study is to evaluate the outcome of body first approach in difficult cases and cases with obscure Calot's triangle in (LC) and to evaluate its feasibility and safety in (LC).

ELIGIBILITY:
Inclusion Criteria:

- All adult patients aging above 18 years old fit for (LC), who presented with symptomatic gall stones by clinical examination and detected by preoperative imaging and intra-operatively have obscure Calot's triangle.

Exclusion Criteria:

* unfit patients.
* Patients with calcular obstructive jaundice.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients aging above 18 years old fit for (LC), who presented with symptomatic gall stones by clinical examination and detected by preoperative imaging and intra-operatively have obscure Calot's triangle.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Safe laparoscopic cholecystectomy. | Baseline
  To achieve critical view of safety during lap cholecystectomy

SECONDARY OUTCOMES:
Evaluation of the body first approach technique | Baseline
  evaluate the body first approach on the rate of conversion to open technique & VBI in patients with obscure calot's triangle.

REFERENCES:
- See also: Laparoscopic cholecystectomy: semi-top-down technique — https://ales.amegroups.org/article/view/5242/html
- See also: Postoperative analgesic effect of ultrasound-guided rectus sheath block and local anesthetic infiltration after laparoscopic cholecystectomy: Results of a prospective randomized controlled trial — http://pubmed.ncbi.nlm.nih.gov/34159732/
- See also: Application of a novel surgical difficulty grading system during laparoscopic cholecystectomy — http://pubmed.ncbi.nlm.nih.gov/34748289/
- See also: Randomized controlled trial comparing the effects of usual gas release, active aspiration, and passive-valve release on abdominal distension in patients who have undergone laparoscopic cholecystectomy — http://pubmed.ncbi.nlm.nih.gov/29266752/
- See also: Body-first approach of laparoscopic cholecystectomy for minimizing vasculobiliary injury: Initial experience — http://pubmed.ncbi.nlm.nih.gov/36650019/
- See also: Laparoscopic Cholecystectomy — http://www.ncbi.nlm.nih.gov/books/NBK448145/
- See also: A three-step conceptual roadmap for avoiding bile duct injury in laparoscopic cholecystectomy: an invited perspective review — http://pubmed.ncbi.nlm.nih.gov/30828991/